CLINICAL TRIAL: NCT00846599
Title: Postprandial Endothelial Dysfunction After a High-Fat Meal in HIV-infected Men
Acronym: PERTH
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Alexandra Mangili, MD, MPH, Tufts University School of Medicine
Other Study IDs: SUB730
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection; Cardiovascular Risk; HIV Infections
Keywords: brachial artery ultrasound; brachial artery reactivity; HIV; human immunodeficiency virus; cardiovascular risk; omega three; saturated fat; sustiva; atripla; kaletra; treatment naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: High omega-3
  Interventions: Other: Omega-3 study meal
- 2: High saturated fat
  Interventions: Other: Saturated fat study meal

INTERVENTIONS:
Other: Omega-3 study meal — Participant will eat a study meal high in omega-3 fatty acids.
  Groups: 1
Other: Saturated fat study meal — Participant will eat a study meal high in saturated fat.
  Groups: 2

SUMMARY:
The purpose of this study is to examine the postprandial (anytime after a meal) effect of different dietary fats on endothelial function in HIV-infected and HIV-uninfected men.

DETAILED DESCRIPTION:
This study requires two visits. Once determined eligible by the study criteria, during the first visit the participant will be randomly placed to receive one of two high-fat meals. The participant will receive the other study meal during the second visit. At each visit, brachial artery ultrasounds will be performed before and 3 hours after the meal is eaten. The sample size is 50 subjects. This study will be conducted at the Clinical Research Center at Tufts Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive white male aged >18 years
* Under one of the following treatment categories:

  * Treatment naive or have never taken any HIV medications
  * Taking Kaletra
  * Taking Sustiva
  * Taking Atripla

Exclusion Criteria:

* Smoker
* Pre-existing diagnosis or treatment for the following:

  * Lipid disorder
  * Cardiovascular disease
  * High blood pressure
  * Diabetes
* Acute opportunistic infection or malignancy within last 3 months or current therapy for either
* Active IV drug use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected white males who have identified themselves with concerns about diet or cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To measure flow-mediated dilation before and after eating the two study meals. | Study visit 1 and 2

SECONDARY OUTCOMES:
To compare the effect of different dietary fats on endothelial function. | Study visit 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Mangili, MD, MPH, Principal Investigator — Tufts University School of Medicine
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- See also: PERTH Study — http://www.tufts.edu/med/nutrition-infection/research/dom/study-perth.html